CLINICAL TRIAL: NCT00499174
Title: A Phase III Study of Active Surveillance Therapy Against Radical Treatment in Patients Diagnosed With Favourable Risk Prostate Cancer [START]
Brief Title: Observation or Radical Treatment in Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not meeting accrual target.
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); Radiation Therapy Oncology Group (Network); Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR11; U10CA077202 (NIH); CAN-NCIC-CTG-PR11 (Registry Identifier: PDQ); CALGB-140602 (Other: CALGB Assigned Trial Code); SWOG-PR11 (Other: SWOG Assigned Trial Code); CDR0000557348 (Other: PDQ); RTOG-0873 (Other: RTOG); ECOG-JPR.11 (Other: ECOG Assigned Trial Code); ICR-CTSU-ProSTART (Other: CTSU)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
Keywords: stage II prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Surveillance (No Intervention): Active surveillance with radical intervention at the time one or more of the following occur: Biochemical progression; Grade progression; Clinical progression
- Radical Intervention (Active Comparator): Radical prostatectomy or radiotherapy based on patient and physician preference
  Interventions: Procedure: conventional surgery; Radiation: brachytherapy; Radiation: external beam radiation therapy; Procedure: Biopsies

INTERVENTIONS:
Procedure: conventional surgery — Radical prostatectomy
  Arms: Radical Intervention
Radiation: brachytherapy — high dose rate temporary seed implant; permanent seed implant.
  Arms: Radical Intervention
Radiation: external beam radiation therapy — 3D conformal radiation therapy; intensity modulated radiation therapy.
  Arms: Radical Intervention
Procedure: Biopsies — Periodic repeat biopsies
  Arms: Radical Intervention

SUMMARY:
RATIONALE: Sometimes prostate tumours may not need treatment until they progress. In this case, observation may be sufficient. Radical treatments, such as radical prostatectomy or radiation therapy, may be effective in treating prostate cancer when it is first diagnosed. It is not yet known whether active surveillance is more effective than radical treatment as an initial intervention in favorable prognosis prostate cancer.

PURPOSE: This randomized phase III trial is studying active surveillance to see how well it works compared with radical treatment as an initial intervention in patients with favorable prognosis prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare disease-specific survival of patients with favorable risk prostate cancer treated with radical prostatectomy or radical radiotherapy at the time of initial diagnosis vs active surveillance and selective intervention based on pre-specified biochemical, histological, or clinical progression criteria.

Secondary

* To compare overall survival, quality of life using the EPIC-26, RAND SF-12, and State-Trait Anxiety Inventory, distant disease-free survival, PSA relapse/progression after radical intervention, and initiation of androgen deprivation therapy between the two treatment arms.
* To determine the proportion of patients on the active surveillance arm who receive radical intervention for prostate cancer.
* To determine if PSA doubling-time prior to diagnosis predicts eventual outcome.
* To determine if molecular biomarkers predict outcome.

OUTLINE: This is a prospective, randomized, multicenter study. Patients are stratified by treatment center, ECOG performance status (0 vs 1 or 2), disease stage (T1 vs T2), baseline PSA value (ng/mL or μg/L) (< 5.0 vs ≥ 5.0 and ≤ 10.0), and age (< 65 years vs ≥ 65 years). Patients are randomized to 1 of 2 arms.

* Arm I: Patients undergo radical intervention (radical prostatectomy or radiotherapy [external-beam radiotherapy 5 days a week for 4-8 weeks; permanent prostate brachytherapy; or high-dose rate temporary brachytherapy], based on patient and physician preference).
* Arm II: Patients undergo active surveillance with radical intervention at the time one or more pre-specified criteria (biochemical progression, histologic/grade progression, and/or clinical progression) are met.

Quality of life is assessed by the EPIC-26, RAND SF-12, and State Anxiety Inventory at baseline, periodically during study treatment, and after completion of radical treatment.

After completion of radical treatment, patients are followed every 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Diagnosed within 6 months prior to randomization
* Patient has been classified as favorable risk as defined by the following:

  * Clinical stage T1b, T1c, T2a, or T2b at the time of diagnosis
  * Clinical (diagnostic biopsy) Gleason score ≤ 6
  * PSA ≤ 10.0 ng/mL
* Physical examination, rectal examination, and transrectal ultrasound have been done within 6 months prior to randomization and radiographic studies, if indicated, are negative for metastasis
* Patient is a suitable candidate for radical prostatectomy or radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0, 1, or 2
* Patient has a minimum life expectancy of > 10 years
* In centers participating in the quality of life component of the study, the patient is able (i.e., sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French
* No history of other malignancies, except adequately treated non-melanoma skin cancer, adequately treated superficial bladder cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years from study randomization

PRIOR CONCURRENT THERAPY:

* No previous treatment for prostate cancer, including surgery (excluding biopsy and TURP), radiotherapy, or androgen deprivation therapy for greater than 3 months
* No planned androgen therapy except in the context of radical therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-12-06 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2013-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence H. Klotz, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Adam S. Kibel, MD, Study Chair — Washington University Siteman Cancer Center; Martin G. Sanda, MD, Study Chair — Beth Israel Deaconess Medical Center; Ian M. Thompson, MD, Study Chair — The University of Texas Health Science Center at San Antonio; Richard Choo, M.D, Study Chair — Mayo Clinic; Chris Parker, M.D, Study Chair — Royal Marsden Hospital, Sulton, UK
Locations (13):
- Canada (13):
  - Clinical Research Unit at Vancouver Coastal, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fung-Kee-Fung SD, Porten SP, Meng MV, Kuettel M. The role of active surveillance in the management of prostate cancer. J Natl Compr Canc Netw. 2013 Feb 1;11(2):183-7. doi: 10.6004/jnccn.2013.0026. PMID 23411385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Surveillance | Radical Intervention
Started | 78 | 102
Completed | 0 | 93
Not Completed | 78 | 9
Not completed — Physician Decision | 78 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Surveillance | Radical Intervention | Total
Number analyzed (Participants) | 78 | 102 | 180
Age, Customized [Number; unit: years]
  age group : 40-49 | 0 | 2 | 2
  age group : 50-59 | 9 | 22 | 31
  age group : 60-69 | 48 | 56 | 104
  age group : >= 70 | 21 | 20 | 41
  age group : Missing | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 78 | 102 | 180
Disease Stage* [Number; unit: participants] — *According to the 6th Edition of the TNM Classification of Malignant Tumours. T1b Tumour incidental histological finding in more than 5% of tissue resected; T1c Tumour identified by needle biopsy, e.g., because of elevated prostate-specific antigen (PSA); T2a Tumour involves one-half of one lobe or less. T2b Tumour involves more than one-half of one lobe, but not both lobes.
  participants
    T1B | 1 | 0 | 1
    T1C | 64 | 79 | 143
    T2A | 12 | 20 | 32
    T2B | 1 | 3 | 4
ECOG Performance Status* [Number; unit: participants] — *ECOG PERFORMANCE STATUS 0 : Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  participants
    0 | 73 | 98 | 171
    1 | 5 | 4 | 9
PSA value [Number; unit: participants]
  < 5. ug/L | 43 | 55 | 98
  >= 5. ug/L | 35 | 47 | 82
Gleason Score (Combined)* [Count of Participants; unit: Participants] — *Gleason score: A grading system for prostate carcinoma devised by Dr. Donald Gleason in 1977 as a method for predicting the behavior of prostate cance.
  ≤ 6: cancer cells that look similar to normal cells and suggest cancer grow slowly.
  7: intermediate risk for aggressive cancer. 8 - 10: cancers spread more rapidly, these cancers are often referred to as poorly differentiated or high grade.
  Participants
    6 | 78 | 102 | 180
    Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-specific Survival
Description: Time from the date of randomization to the date of death due to prostate cancer.
Time Frame: 5 years 6 months
Population: Due to difficulty in accruing patients to the trial, the trial was closed early, there is no patient died of prostate cancer. Thus, no analysis was done.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Radical Intervention | Active Surveillance
Number analyzed (Participants) | 78 | 102
years | NA [NA to NA] — There is no patient died of prostate cancer reported in the trial, so none of the reported value is available. | NA [NA to NA] — There is no patient died of prostate cancer reported in the trial, so none of the reported value is available.

2. Secondary Outcome: Overall Survival
Description: Time from randomization to the date of death due to any causes.
Time Frame: 5 years 6 months
Population: Due to lower patients accrual rate, the trial was closed early with only 3 events reported in the trial, Thus.no formal analysis had been done.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Active Surveillance | Radical Intervention
Number analyzed (Participants) | 78 | 102
years | NA [NA to NA] — There is no patient died of prostate cancer reported in the trial, so none of the reported value is available. | NA [NA to NA] — There is no patient died of prostate cancer reported in the trial, so none of the reported value is available.

ADVERSE EVENTS:
Time Frame: q 3 months for 2 years then every 6 months for 5 years and 6 months.
Description: Adverse events graded according to CTCAE V4.0
Arm/Group | Active Surveillance | Radical Intervention
All-Cause Mortality (participants affected / at risk) | 1/78 | 2/99
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/99
Other Adverse Events (participants affected / at risk) | 57/78 | 65/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Surveillance (N=78) | Radical Intervention (N=99)
Fatigue (General disorders) | 15 (15) | 7 (7)
Pain Testicle (General disorders) | 1 (1) | 9 (9)
Incontinence, urinary (Renal and urinary disorders) | 3 (3) | 11 (11)
Urinary frequency (Renal and urinary disorders) | 34 (34) | 29 (29)
Urinary retention (Renal and urinary disorders) | 12 (12) | 12 (12)
Ejaculatory dysfunction (Reproductive system and breast disorders) | 37 (37) | 41 (41)

LIMITATIONS AND CAVEATS:
Due to the early termination of the trial, the small number of patients and the shorter follow up, the reported information may not be reliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No